CLINICAL TRIAL: NCT06031571
Title: Effect of Dry Cupping Massage Versus Myofascial Release Therapy in Patients With Mechanical Non-specific Neck Pain: a Quasi-experimental Study
Brief Title: Effect of Dynamic Cupping Versus Myofascial Release Therapy in Patients With Mechanical Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal Abouelyazeed Ali, Lecturer of Physical Therapy for Women's Health, South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: cupping vs release
Record Dates: First submitted 2023-08-27; First posted 2023-09-11 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Mechanical Neck Pain

STUDY DESIGN:
Intervention Model Description: 38 participants will be assigned at random into 2 equal groups: group A (will receive dry cupping massage technique in addition to traditional exercises for 3 sessions per week for 12 sessions), and group B (will receive myofascial release technique in addition to traditional exercises for 3 sessions per week for 12 sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): group A (will receive cupping massage technique in addition to traditional exercises)
  Interventions: Procedure: dry cupping massage
- Group B (Experimental): group B (will receive myofascial release technique in addition to traditional exercises)
  Interventions: Procedure: Myofacial release

INTERVENTIONS:
Procedure: dry cupping massage — Dry cupping is a form of massage therapy that involves using Hijamat cups without skin injury while applying suction and then performing circular and transverse movements
  Other Names: traditional exercises (neck stretching and strengthening exercises)
  Arms: group A
Procedure: Myofacial release — Myofascial release is a form of manual therapy using hands-on techniques to regain tissue extensibility and elasticity
  Other Names: traditional exercises (neck stretching and strengthening exercises)
  Arms: Group B

SUMMARY:
A Quasi-experimental study will investigate the effect of dry cupping massage versus myofascial release on patients with mechanical neck pain.

DETAILED DESCRIPTION:
PURPOSE: To investigate the effect of dry cupping massage versus myofascial release on pain level, range of motion, and functional level in mechanical neck pain…

BACKGROUND: Neck pain is a multivariate disease and is a leading issue in a modernized society. The economic burden of neck pain is remarkable and includes treatment costs, reduced productivity, and job-related problems (Cohen, 2015).

There is no one definitive treatment for neck pain. However, different pharmacological and non-pharmacological treatments have been recommended, including laser therapy, massage, acupuncture, yoga, and aquatic therapy (Corvillo et al., 2020). However, no studies are focusing on comparing the effect of dynamic cupping and myofascial release in mechanical neck pain.

HYPOTHESES: There will be a non-significant difference between dry cupping massage and myofascial release on pain level, range of motion, and functional level in patients with mechanical neck pain…

RESEARCH QUESTION: Will there be a difference between dry cupping massage versus myofascial release on pain level, range of motion, and functional level in patients with mechanical neck pain?

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18- 40 years.
2. Participants have experienced mechanical neck pain for at least the previous 3 months.

Exclusion Criteria:

* Participants aged below 18 years-old and those above 40 years old
* Mechanical neck pain due to trauma, disc protrusion, congenital deformity of the spine, spinal stenosis, and rheumatoid disease.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-07-12 (Estimated); Study Completion 2024-07-20 (Estimated)

PRIMARY OUTCOMES:
Cervical range of motion | Assessment will be done pre and post treatment sessions (3 sessions/week, total of 12 sessions in 4 weeks)
  Cervical flexion and extension ranges of motion are measured by goniometer in numerical degrees

SECONDARY OUTCOMES:
Neck Disability index | Assessment will be done pre and post treatment sessions (3 sessions/week, total of 12 sessions in 4 weeks)
  The neck disability index is a questionnaire has been designed to inform how neck pain has affected different aspects in everyday life.
Visual analog scale | Assessment will be done pre and post treatment sessions (3 sessions/week, total of 12 sessions in 4 weeks)
  The visual analog scale is a scale for pain severity assessment with range from 0 (o pain) to 10 (intolerable pain)

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of physical therapy, South Valley University, Qina, Qena Governorate
  - Faculty of physical therapy, Cairo